CLINICAL TRIAL: NCT04506918
Title: Comparison of Short Message Service (SMS) and Interactive Voice Response (IVR) Mobile Phone Surveys for Non-communicable Disease Risk Factor Surveillance in Tanzania
Brief Title: Comparison of SMS and IVR Surveys in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318 - abc
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; interactive voice response; short message service
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two arms : 1) IVR or 2) SMS. Participants in the first study arm will receive an IVR survey. Participants in the second study arm will receive a SMS survey.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVR survey (Experimental): Participants will receive an IVR survey
  Interventions: Other: IVR survey
- SMS survey (Experimental): Participants will receive an SMS survey
  Interventions: Other: SMS survey

INTERVENTIONS:
Other: IVR survey — Participants will receive an IVR survey
  Arms: IVR survey
Other: SMS survey — Participants will receive a SMS survey
  Arms: SMS survey

SUMMARY:
This study focuses on mechanisms to adapt the performance of interactive voice response (IVR) and short message service (SMS) surveys conducted in low-and middle-income (LMIC) setting (Tanzania) and evaluates how the two survey modalities (IVR and SMS) affect survey metrics, including response, completion and attrition rates.

DETAILED DESCRIPTION:
Using random digit dialing (RDD) sampling technique, participants will be randomized to one of two arms : 1) IVR or 2) SMS. Participants in the first study arm will receive an IVR survey. Participants in the second study arm will receive a SMS survey. The IVR and SMS questionnaires contain a set of demographic questions and one non-communicable disease (NCD) module (alcohol, or tobacco, or diet, or physical activity, or blood pressure and diabetes). We will examine contact, response, refusal and cooperation rates and demographic representativeness by each study arm.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* Conversant in the Swahili language

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6483 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Cooperation Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, cooperation rate is defined as I/(I+P+R) where I is the number of participants with complete interviews, P is the number of participants with partial interviews, and R is the number of participants with refusals and breakoffs.
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, response rate is defined as (I+P)/(I+P+R+eU) where I is the number of participants with complete interviews, P is the number of participants with partial interviews, R is the number of participants with refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, refusal rate is defined as (R)/(I+P+R+eU) where R is the number of participants with refusals and breakoffs, I is the number of participants with complete interviews, P is the number of participants with partial interviews, and eU is the estimated eligible proportion of unknowns
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, contact rate is defined as (I+P+R)/(I+P+R+eU) where I is the number of participants with complete interviews, P is the number of participants with partial interviews, R is the number of participants with refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Gibson, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; Honorati Masanja, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722